CLINICAL TRIAL: NCT03227263
Title: BABH Study: Efficacy and Safety of Bevacizumab on Severe Bleedings Associated With Hemorrhagic Hereditary Telangiectasia (HHT). A National, Multicenter Phase III Study
Brief Title: BABH Study: Efficacy and Safety of Bevacizumab on Severe Bleedings Associated With Hemorrhagic Hereditary Telangiectasia (HHT).
Acronym: BABH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL17_0018; 2017-001031-39 (EudraCT Number)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2020-06

CONDITIONS: Rendu Osler Disease; Telangiectasia, Hereditary Hemorrhagic
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); VEGF therapy; Bevacizumab
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab (Experimental): Intravenous infusion of Bevacizumab at a dose of 5 mg/kg
  Interventions: Drug: Bevacizumab
- Placebo (Placebo Comparator): 0.9% of sodium chloride is infused every 14 days for 6 consecutive administrations
  Interventions: Drug: sodium chloride 0.9%

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (Avastin®) concentrate at 25mg/mL is diluted at 5 mg/kg for infusion every 14 days for 6 consecutive administrations
  Arms: Bevacizumab
Drug: sodium chloride 0.9% — 0.9% of sodium chloride is infused every 14 days for 6 consecutive administrations
  Arms: Placebo

SUMMARY:
The recognized manifestations of HHT are all due to abnormalities of vascular structure. Epistaxis and digestive arteriovenous malformations may be responsible for severe hemorrhages in 5% of HHT patients, requiring repeated blood transfusions and are associated with high morbidity. There is currently no standard and efficient management of this severe symptom. It is also well known that HHT-associated hemorrhages have the greatest negative impact on quality of life among HHT patients, and is responsible for anemia, blood transfusions, hospitalizations, depressive syndrome and a high psycho-social impact.

Since 2006, it has been suggested by animal models and then by clinical reports that anti-VEGF therapy may be useful to treat HHT. 4 case reports have been published on efficacy of intravenous bevacizumab, a humanized monoclonal antibody in HHT on severe hemorrhages.

Intravenous bevacizumab has been used in a previous clinical trial to measure efficacy and tolerance of this drug in HHT patients with severe liver involvement. Furthermore, a reduction was observed in the duration of the nosebleeds after treatment and was encouraging to treat bleeding. We completed this study by a pharmacokinetic-pharmacodynamic (PK-PD) model in order to assess the individual concentration-effect relationship of bevacizumab.

However, no randomized prospective study has been performed and published to evaluate the efficacy in this indication. A total of 24 patients will be randomized versus placebo in a multicenter phase III trial. The Avastin or placebo will be infused at 5mg/kg every 14 days with a total of 6 cures with a 3 months following period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who have given their free informed and signed consent.
* Patients affiliated to a social security scheme or similar.
* Patients monitored for clinically confirmed HHT (presence of at least three Curaçao criteria) and / or with molecular biology confirmation.
* Blood transfusions with the requirement for at least 4 units of blood in the 3-month period before study enrollment, related to epistaxis or digestive bleeding.

Exclusion Criteria:

* Women who are pregnant or nursing (lactating), women of child-bearing potential without reliable contraception during the treatment and for at least 6 months after the last dose.
* Patients who are protected adults under the terms of the law (French Public Health Code).
* Refusal to consent.
* Patients for whom the diagnosis of HHT has not been confirmed clinically and / or by molecular biology study.
* Active infection and/or fever>38°C
* Participation in another clinical trial within 28 days prior to inclusion.
* Hypersensitivity to the active substance or to any of the excipients.
* Known hypersensitivity to products of Chinese hamster ovary cells (CHO) or other recombinant human or humanized antibodies.
* Patients who have taken Avastin ® intravenously in the 6 months prior to inclusion.
* Patients who have had a therapeutic endoscopy for gastrointestinal bleeding or ENT surgery for epistaxis will have to wait at least 3 months less after treatment to be included if bleeding persists.
* Patients who had a surgery in the month prior inclusion or planned surgery within 6 months
* Severe peripheral arterial disease with ulcerations
* Unhealed wound
* Thrombosis in the 6 months prior to inclusion
* Anticoagulant treatment
* Uncontrolled high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
number of red blood cell transfusions | 6 months

SECONDARY OUTCOMES:
hemoglobin | 3 months
  The relative evolution in hemoglobin level at 3 months after the beginning of the treatment is compared to the value measured at inclusion
hemoglobin | 6 months
  The relative evolution in hemoglobin level at 6 months after the beginning of the treatment is compared to the value measured at inclusion
epistaxis frequency | 3 months before treatment up to 6 months from the inclusion
  Comparison of an average over a 3-month period before and after the treatment.
duration of nosebleeds | 3 months before treatment up to 6 months from the inclusion
  Comparison of an average over a 3-month period before and after the treatment.
digestive vascular malformations | 6 months
  Comparison of digestive endoscopy before and after treatment if gastrointestinal bleeding have already externalized before treatment
quality of life (SF36). | 3 months
  Comparison of SF36 questionnaire before and after treatment.
quality of life (SF36). | 6 months
  Comparison of SF36 questionnaire before and after treatment.
severity epistaxis score (ESS). | 3 months
  Comparison of ESS questionnaire before and after treatment
severity epistaxis score (ESS). | 6 months.
  Comparison of ESS questionnaire before and after treatment
To evaluate pharmacokinetics of bevacizumab dose | Before each 6 infusions
  Description of bevacizumab serum concentrations over time, the relationship between bevacizumab concentrations and adverse events and clinical/biological endpoints
To evaluate pharmacokinetics of bevacizumab dose | 2 hours after the first treatment infusion
  Description of bevacizumab serum concentrations over time, the relationship between bevacizumab concentrations and adverse events and clinical/biological endpoints
adverse events | up to 6 months
  To assess the safety of bevacizumab.Tolerance will be evaluated by recording adverse events and by clinical examinations during the treatment period and the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: DUPUIS-GIROD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - CHU d'Angers, Angers
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Femme Mère Enfant, Bron
  - CHU de Montpellier Hôpital St Eloi, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dupuis-Girod S, Riviere S, Lavigne C, Fargeton AE, Gilbert-Dussardier B, Grobost V, Leguy-Seguin V, Maillard H, Mohamed S, Decullier E, Roux A, Bernard L, Saurin JC, Saroul N, Faure F, Cartier C, Altwegg R, Laccourreye L, Oberti F, Beaudoin M, Dhelens C, Desvignes C, Azzopardi N, Paintaud G, Hermann R, Chinet T. Efficacy and safety of intravenous bevacizumab on severe bleeding associated with hemorrhagic hereditary telangiectasia: A national, randomized multicenter trial. J Intern Med. 2023 Dec;294(6):761-774. doi: 10.1111/joim.13714. Epub 2023 Aug 23. PMID 37592715